CLINICAL TRIAL: NCT05940870
Title: A Prospective, Open-label, Post-marketing Observational Study Assessing the Safety and Efficacy of Nerivio for Migraine Prevention in Real-world Environment.
Brief Title: A Prospective Post-marketing Observational Study Assessing the Safety and Efficacy of Nerivio for Migraine Prevention.
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: TCH015
Record Dates: First submitted 2023-06-28; First posted 2023-07-11 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2023-06

CONDITIONS: Migraine
Keywords: migraine prevention; Remote electrical neuromodulation
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Nerivio treatment for migraine prevention: Patients with migraine who recieved the Nerivio device for migraine prevention therapy
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — Patients with migraine who received the Nerivio device for migraine prevention therapy

SUMMARY:
Nerivio is a remote electrical neuromodulation (REN) device that is FDA-cleared for migraine prevention (as well as for acute treatment of migraine), in individuals 12 and older. The study is a post-marketing, observational, prospective, real-world evidence study assessing the safety, efficacy, and health economics outcomes of Nerivio for migraine prevention in a real-world environment. The study population is naïve Nerivio users, aged 12 and up, who were prescribed Nerivio by their healthcare provider for either prevention treatment (for use every other day) or dual-use treatment (for use every other day and upon the onset of a migraine). The study period per participant is six months. During this period, participants will be requested to use Nerivio according to the instructions of their healthcare provider and to fill out a short daily questionnaire in the Nerivio application

DETAILED DESCRIPTION:
Nerivio is an FDA-approved remote electrical neuromodulation (REN) device for the acute and/or preventive treatment of migraine with or without aura. Nerivio delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application. The study will assess the safety and efficacy of Nerivio, used every other day for prevention and possibly whenever needed for acute treatment, as prescribed to participants by their own healthcare provider. The study will also assess certain health economics outcomes related to the treatment.

Patients aged 12 or above who were prescribed Nerivio for prevention or dual-use treatment of migraine after April 1st.

New Nerivio users will be sent an invitation message (via in-app notification and email), inviting them to fill out a Screening Eligibility Questionnaire. Those who meet the eligibility criteria will be offered to participate in the study. Candidate participants will then complete and sign an electronic Informed Consent Form (ICF). Immediately following this, participants will receive a Baseline Questionnaire with questions relating to the time period prior to using Nerivio.

The study duration for each participant is 24 weeks. During this time, participants will fill out the Daily Diary in the Nerivio App. In the middle of the study period (end of week 12), and at the end of the 24 weeks, participants will be asked to fill out follow-up questionnaires (Mid-study questionnaire & Completion questionnaire) with questions on migraine and related symptoms, medication intake, health economics, and satisfaction with the treatment.

Participants who stop treatment will be sent a Completion questionnaire concerning the reason for their withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years old or above.
* Were prescribed with Nerivio for prevention (or for dual use) after April 1st.
* Have performed up to 3 preventive treatment sessions and have never used Nerivio before that.
* Have had at least 4 migraine attacks per month (according to self-report).
* Stable on the same migraine prevention treatment for the last two months prior to enrollment.
* Signed an electronic Informed Consent Form and agreed to fill the Daily Diary in the Nerivio mobile app on a daily basis.

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Migraine patients aged 12 or above who were prescribed Nerivio for prevention or dual use treatment of migraine
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in monthly mean number of migraine days from baseline to weeks 9-12 of the study. | 12 weeks
  Change in number of monthly migraine days depicting the change in the number of migraine days from baseline, as reported by the patient, to weeks 9-12 of the study.
  Migraine Day: a calendar day with a headache that is either accompanied by at least one of the following symptoms: 1. Photophobia/phonophobia 2. nausea (with or without vomiting), OR is treated with a migraine-specific acute medication.
Rate of Adverse Events (Safety and Tolerability) | 24 weeks
  Numer of AE, SAE and Device-related Adverse Events

SECONDARY OUTCOMES:
Change in the monthly number of monthly headache days from weeks 1-4 to weeks 9-12. | 12 weeks
  Change in number of monthly headache days depicting the change in the number of headache days from weeks 1-4 to weeks 9-12.
  Headache Day: a calendar day with a headache of any severity.
Change in monthly mean number of migraine days from baseline to weeks 21-24 | 24 weeks
  Change in number of monthly migraine days depicting the change in the number of migraine days from baseline, as reported by the patient, to weeks 21-24 of the study.
Change in the monthly mean number of prescription acute medication days from weeks 1-4 to weeks 9-12. | 12 weeks
  Change in number of monthly prescribed acute medication intake days depicting the change in the number of prescribed acute medication intake days from weeks 1-4 to that of weeks 9-12 of the study
  Acute Medication Day: a calendar day on which the participant took at least one prescribed medication for acute treatment of migraine.

OTHER OUTCOMES:
Change in the number of monthly headache days from weeks 1-4 to weeks 21-24. | 24 weeks
  Change in number of monthly headache days depicting the change in the number of headache days from weeks 1-4 to weeks 21-24
Change in the monthly mean number of prescription acute medication days from weeks 1-4 to weeks 21-24. | 24 weeks
  Change in number of monthly prescribed acute medication intake days depicting the change in the number of prescribed acute medication intake days from weeks 1-4 to that of weeks 21-24 of the study
Change in monthly mean number of migraine days from baseline to weeks 21-24 of the study. | 24 weeks
  Change in number of monthly migraine days depicting the change in the number of migraine days from baseline, as reported by the patient, to weeks 21-24 of the study.
Change in the monthly mean number of presenteeism days during the study. | 24 weeks
  Change in number of monthly presenteeism days depicting the change in the number of presenteeism days from weeks 1-4 to that of the subsequent study months.
  Presenteeism Day: a calendar day on which the participant is at work (or school) with the presence of moderate/severe functional disability
Change in the monthly mean number of absenteeism days during the study | 24 weeks
  Change in number of monthly absenteeism days depicting the change in the number of absenteeism days from weeks 1-4 to that of the subsequent study months.
  Absenteeism Day: a calendar day on which the participant is absent from work (or school) due to migraine disability.
Adherence to treatment | 24 weeks
  Proportion of participants (in percent) treating, on average, at least 10 times per 4-weeks period during the study.
Change in the Patient Global Impression of Severity from baseline to the end of weeks 2 and 24 | 24 weeks
  Change in the Patient's Global Impression of Severity (PGI-S) from baseline to the end of weeks 12 and 24.
  Patient's Global Impression of Severity score scale is a Scale text (single-question scale): Since the start of the study, my overall status is:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Change in the Patient Global Impression of Change from baseline to the end of weeks 2 and 24 | 24 weeks
  hange in the Patient's Global Impression of Change(PGI-G) from baseline to the end of weeks 12 and 24.
Self report of tolerability | 24 weeks
  Change in the Patient's Self report of tolerability during the study period This outcome measure is a single-item self-report scale to assess the patient's subjective experience of the extent to which the treatment was well-tolerated.
  Scale text: To what extent was the treatment well tolerated?
  1. Completely tolerable
  2. Very tolerable
  3. Moderately tolerable
  4. Slightly tolerable
  5. Not at all tolerable
Prediction of a migraine day | 24 weeks
  prediction of a migraine day based on prodromal symptoms. Predictive accuracy, measured as the difference between the observed values and predicted values of the occurrence of a migraine day in the following (predicted) day.

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark Inbar, Principal Investigator — Theranica
Locations (1):
- Theranica Inc USA, Bridgewater, New Jersey, United States